CLINICAL TRIAL: NCT05174949
Title: Targeted HD-tDCS for Reducing Post-stroke Movement Impairments
Brief Title: Targeted High-definition Transcranial Direct Current Stimulation (HD-tDCS) for Reducing Post-stroke Movement Impairments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma Shared Clinical and Translational Resources (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 14011
Record Dates: First submitted 2021-11-09; First posted 2022-01-03 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: Stroke; upper limb impairment; HD-tDCS
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This sham-controlled cross-over study design will include three visits: 1) anodal stimulation targeting ipsilesional primary motor cortex, 2) cathodal one at the contralesional premotor cortex, 3) a sham stimulation visit. The sequence of the stimulations will be randomized and double-blinded. After each intervention, there will be at least 2 weeks wash-out period before participants receive the next intervention and assessments.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sham, Anodal, Cathodal (Experimental): Treatment order 1: Sham, Anodal, Cathodal
  Interventions: Device: Transcranial direct current stimulation (high-definition)
- Anodal, Cathodal, Sham (Experimental): Treatment order 2: Anodal, Cathodal, Sham
  Interventions: Device: Transcranial direct current stimulation (high-definition)
- Cathodal, Sham, Anodal (Experimental): Treatment order 3: Cathodal, Sham, Anodal
  Interventions: Device: Transcranial direct current stimulation (high-definition)
- Sham, Cathodal, Anodal (Experimental): Treatment order 4: Sham, Cathodal, Anodal
  Interventions: Device: Transcranial direct current stimulation (high-definition)
- Cathodal, Anodal, Sham (Experimental): Treatment order 5: Cathodal, Anodal, Sham
  Interventions: Device: Transcranial direct current stimulation (high-definition)
- Anodal, Sham, Cathodal (Experimental): Treatment order 6: Anodal, Sham, Cathodal
  Interventions: Device: Transcranial direct current stimulation (high-definition)

INTERVENTIONS:
Device: Transcranial direct current stimulation (high-definition) — Three conditions (2 mA, 20 mins):
  1. anodal stimulation over the ipsilesional primary motor cortex
  2. cathodal one over the contralesional premotor cortex
  3. Sham

SUMMARY:
Stroke is the leading cause of serious, long-term disability. The emergence of abnormal muscle synergies following a stroke presents a major limitation to the recovery of independent function. Despite the development of many interventions for movement recovery post-stroke, rehabilitation treatments are minimally effective to the muscle synergy impairment. Previous studies have found that muscle synergy impairment is associated with the damage to the corticospinal tract and the maladaptive recruitment of the contralesional cortico-reticulospinal tract. The investigators hypothesize that facilitating the damaged cortico-spinal tract (via primary motor cortex) and/or inhibiting the contralesional cortico-reticulospinal tract (via dorsal premotor cortex) will reduce muscle synergy impairment. In this pilot project, the investigators propose to run a proof-of-concept pilot trial to evaluate the effect of the targeted high-definition transcranial direct current stimulation (HD-tDCS) on mitigating muscle synergy impairment.

DETAILED DESCRIPTION:
This randomized, double-blinded, sham-controlled cross-over study will include three stimulation conditions: 1) anodal stimulation over the ipsilesional primary motor cortex, 2) cathodal one over the contralesional premotor cortex, 3) sham stimulation in chronic hemiparetic stroke patients.

Stroke participants (> 3 months after stroke) with moderate to severe motor impairments (Fugl-Meyer Motor Assessment - Upper Extremity score between 10-40, in absence of clinically defined sensory deficits) and an ischemic unilateral subcortical lesion will receive each type of stimulation for 20 minutes.

Their brain activity and behavior data will be collected for the outcome measures.

The patient time commitment in this study is approximately 7 weeks where subjects have 3 x 1-day intervention and measurements, with 2 weeks washout period in between.

The total number of potential enrolled subjects in this pilot study is 12.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic unilateral stroke lesion (confirmed by the most recent clinical or radiological reports) at least 3 months prior to participation in this project.
* Paresis confined to one side, with moderate to severe motor impairment of the upper limb (Fugl-Meyer upper extremity scores of 10-40)
* Capacity to provide informed consent

Exclusion Criteria:

* Muscle tone abnormalities and motor or sensory impairment in the unimpaired limb
* Severe wasting or contracture or significant sensory deficits in the paretic upper limb
* Severe cognitive or affective dysfunction that prevents normal communication and understanding of consent or instruction
* Severe concurrent medical problems (e.g. cardiorespiratory impairment)
* Using a pacemaker
* Metal implants in the head
* Known adverse reaction to TMS and tDCS
* Pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing the value of research and furthering the advancement of public knowledge. We recognize that the public dissemination of our scientific results can facilitate the creation of collaborative efforts with domestic and international collaborators. Furthermore, we recognize that the proposed project may result in novel ideas for new methods, technologies, and data that could benefit the entire research community. Therefore, final research data will be shared openly and timely in accordance with the most recent NIH guidelines (http://grants.nih.gov/grants/policy/data_sharing/) while being mindful that the confidentiality and privacy of participants in research must be protected at all times.

REFERENCES:
- [Result] Williamson J, James SA, Apple B, Sharps J, Sidorov E.V., Yang Y, (2022), High Definition Transcranial Direct Current Stimulation for Improving Upper Extremity Motor Function post Stroke. June 8-10, the 3rd International Workshop on Non-Invasive Brain Stimulation (NIBS) 2022.
- [Result] Lepak L.V., Cheema C.F, James S.A., Yang Y (2023), Computer-Guided Non-Invasive High-Definition Transcranial Direct Current Brain Stimulation as a Targeted Intervention after a Stroke, American Physical Therapy Association (APTA) Combined Sections Meeting (CSM), San Diego, CA, Feb 23-25, 2023
- [Derived] Williamson JN, James SA, He D, Li S, Sidorov EV, Yang Y. High-definition transcranial direct current stimulation for upper extremity rehabilitation in moderate-to-severe ischemic stroke: a pilot study. Front Hum Neurosci. 2023 Oct 12;17:1286238. doi: 10.3389/fnhum.2023.1286238. eCollection 2023. PMID 37900725

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Our primary patient resource is from OU Physician Neurology Clinic and Allied Health Clinical Network. We also seek referrals from clinicians in the Oklahoma City areas and recruit stroke survivors residing in these two areas who wish to participate in the study. The recruitment method include doctor referrals and direct contact (if study doctor's patients) via the study doctor. Recruitment period: 1/18/2022-5/12/2023
Pre-assignment Details: Stroke participants will be examined by the study doctor to verify their admissibility to the study based on the inclusion criteria. Participants will then undergo the upper extremity portion of the Fugl-Meyer Motor Assessment, and a structured interview pertaining to the inclusion criteria.
Groups:
- Sham, Anodal, Cathodal: Transcranial direct current stimulation (high-definition): Three conditions (2 mA, 20 mins) with 2-week wash-out period:
  1. sham
  2. anodal stimulation over the ipsilesional primary motor cortex
  3. cathodal one over the contralesional premotor cortex
- Cathodal, Sham, Anodal: Transcranial direct current stimulation (high-definition): Three conditions (2 mA, 20 mins):
  1. cathodal one over the contralesional premotor cortex
  2. sham
  3. anodal stimulation over the ipsilesional primary motor cortex
- Sham, Cathodal, Anodal: Transcranial direct current stimulation (high-definition): Three conditions (2 mA, 20 mins):
  1. sham
  2. cathodal one over the contralesional premotor cortex
  3. anodal stimulation over the ipsilesional primary motor cortex
- Cathodal, Anodal, Sham: Transcranial direct current stimulation (high-definition): Three conditions (2 mA, 20 mins):
  1. cathodal one over the contralesional premotor cortex
  2. anodal stimulation over the ipsilesional primary motor cortex
  3. sham
Period: Overall Study
Arm/Group | Sham, Anodal, Cathodal | Anodal, Cathodal, Sham | Cathodal, Sham, Anodal | Sham, Cathodal, Anodal | Cathodal, Anodal, Sham | Anodal, Sham, Cathodal
Started | 1 | 4 | 1 | 5 | 2 | 1
Per-protocol (PP) Population | 1 | 4 | 1 | 4 | 2 | 1
Completed | 0 | 1 | 1 | 3 | 2 | 1
Not Completed | 1 | 3 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 1 | 2 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline demographics taken from the per-protocol (PP) population; the PP group includes all participants who signed an informed consent, were randomized to a treatment arm, and completed the baseline assessment. There is one subject is loss of follow-up before the baseline assessment, resulting in a total of 13 subjects included in the baseline analysis.
Groups:
- Sham, Anodal, Cathodal: Treatment order 1: Sham, Anodal, Cathodal
  Transcranial direct current stimulation (high-definition): Three conditions (2 mA, 20 mins):
  1. anodal stimulation over the ipsilesional primary motor cortex
  2. cathodal one over the contralesional premotor cortex
  3. Sham
- Anodal, Cathodal, Sham: Treatment order 2: Anodal, Cathodal, Sham
  Transcranial direct current stimulation (high-definition): Three conditions (2 mA, 20 mins):
  1. anodal stimulation over the ipsilesional primary motor cortex
  2. cathodal one over the contralesional premotor cortex
  3. Sham
- Cathodal, Sham, Anodal: Treatment order 3: Cathodal, Sham, Anodal
  Transcranial direct current stimulation (high-definition): Three conditions (2 mA, 20 mins):
  1. anodal stimulation over the ipsilesional primary motor cortex
  2. cathodal one over the contralesional premotor cortex
  3. Sham
- Sham, Cathodal, Anodal: Treatment order 4: Sham, Cathodal, Anodal
  Transcranial direct current stimulation (high-definition): Three conditions (2 mA, 20 mins):
  1. anodal stimulation over the ipsilesional primary motor cortex
  2. cathodal one over the contralesional premotor cortex
  3. Sham
- Cathodal, Anodal, Sham: Treatment order 5: Cathodal, Anodal, Sham
  Transcranial direct current stimulation (high-definition): Three conditions (2 mA, 20 mins):
  1. anodal stimulation over the ipsilesional primary motor cortex
  2. cathodal one over the contralesional premotor cortex
  3. Sham
- Anodal, Sham, Cathodal: Treatment order 6: Anodal, Sham, Cathodal
  Transcranial direct current stimulation (high-definition): Three conditions (2 mA, 20 mins):
  1. anodal stimulation over the ipsilesional primary motor cortex
  2. cathodal one over the contralesional premotor cortex
  3. Sham
- Total: Total of all reporting groups
Arm/Group | Sham, Anodal, Cathodal | Anodal, Cathodal, Sham | Cathodal, Sham, Anodal | Sham, Cathodal, Anodal | Cathodal, Anodal, Sham | Anodal, Sham, Cathodal | Total
Number analyzed (Participants) | 1 | 4 | 1 | 4 | 2 | 1 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (0) | 51.75 (13.18) | 81 (0) | 62.4 (12.95) | 64.5 (10.6) | 67 (0) | 61 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 1 | 0 | 3
  Male | 1 | 4 | 0 | 3 | 1 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 0 | 4 | 1 | 4 | 2 | 1 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 3 | 1 | 4 | 2 | 1 | 12
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 4 | 1 | 4 | 2 | 1 | 13
Subset of Fugl-Meyer Upper Extremity assessment which is mainly related to the muscle synergy [Mean (Standard Deviation); unit: units on a scale] — The Fugl-Meyer Upper Extremity (FM-UE) subset is a component of the Fugl-Meyer Assessment (FM) assessing motor impairment in individuals with stroke or other arm impairments. The (FM-UE) subset focuses on evaluating motor impairment and recovery using movements assessing strength, coordination, sensation, and range of motion of the upper extremity.
  Each item in the FM-UE subset is scored on a scale from 0-2. These are added together, with higher scores indicating better motor function. The FM-UE subset has 33 items for a maximum possible (highest functioning) score of 66.
  units on a scale | 25 (0) | 25 (11.6) | 8 (0) | 17.75 (6.90) | 12.5 (2.12) | 7 (0) | 18.15 (9.47)
Onset Latency of Transcranial magnetic stimulation (TMS)-evoke motor-evoked potentials (MEP) [Mean (Standard Deviation); unit: ms] — The TMS-induced MEP were assessed to determine the ipsilesional corticospinal tract. The paired-pulse TMS was applied at the respective hotspot for the elbow flexor muscle at the paretic arm over the ipsilesional primary motor cortex. The center of the coil was positioned tangentially to the skull. The patient was considered MEP+ if MEPs of any amplitude are observed at a consistent latency on at least 5 out 10 trials. After determining the status of MEP, at least eight more pulses were applied. We calculated average latency across all positive trials to determine the latency of MEP.
  ms | 23.82 (0) | 49.49 (20.10) | 74.48 (0) | 48.50 (9.81) | 62.66 (14.86) | 60.82 (0) | 52.03 (16.83)
Brain symmetry index [Mean (Standard Deviation); unit: Index] — The brain symmetry index is a measure used to quantify the symmetry or asymmetry between the left and right hemispheres of the brain. It was calculated using EEG data from a 3-minute resting state EEG recording. The scale of the index is from -1 to 1, where zero is considered perfect symmetry between hemispheres and values close to -1 and 1 indicate asymmetry.
  Index | -0.091 (0) | 0.007 (0.120) | -0.091 (0) | 0.093 (0.149) | 0.061 (0.009) | -0.439 (0) | -0.015 (0.173)

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Upper Extremity Assessment Part A
Description: The Fugl-Meyer Upper Extremity (FM-UE) subset is a component of the Fugl-Meyer Assessment (FM) assessing motor impairment in individuals with stroke or other arm impairments. The (FM-UE) subset focuses on evaluating motor impairment and recovery using movements assessing strength, coordination, sensation, and range of motion of the upper extremity.
  Each item in the FM-UE subset is scored on a scale from 0-2. These are added together, with higher scores indicating better motor function. The FM-UE subset has 33 items for a maximum possible (highest functioning) score of 66.
Time Frame: The FM-UE assessment is completed before and immediately after (within 30 min range) the intervention. The mean difference is then calculated (Post-Pre intenvention) and recorded for each treatment group (anodal, cathodal, and sham). .
Population: Eight subjects completed the study were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Anodal Stimulation: Anodal stimulation over the ipsilesional primary motor cortex
- Cathodal Stimulation: Cathodal stimulation over the contralesional premotor cortex.
- Sham: Sham stimulation
Arm/Group | Anodal Stimulation | Cathodal Stimulation | Sham
Number analyzed (Participants) | 8 | 8 | 8
score on a scale | 4.13 (4.29) | 5.38 (3.58) | 0.88 (0.99)
Statistical Analysis 1: Comparison: Anodal Stimulation vs Cathodal Stimulation vs Sham; We will report first anode compared to sham and then cathode compared to sham; Test type: Superiority — We performed a linear regression analysis (generalized estimating equations) in which we compared both intervention groups to the sham group and added a time interaction term; p < 0.0001, Generalized Estimating Equations — Anode compared to sham: p = 0.0516 Cathode compared to sham: p <.0001 . Anode change over time compared to sham p=0.0255 Cathode change over time compared to sham p<.0001; Mean Difference (Final Values) = 5.4, 95% CI 2-sided [2.4 to 8.4], Standard Deviation 3.58 — Anode mean change = 4.13 std = 4.29 CLM = 0.5-7.7 Cathode mean change = 5.38 std = 3.58 CLM=2.4-8.4

2. Secondary Outcome: Change in Onset Latency of Transcranial Magnetic Stimulation (TMS)-Evoke Motor-evoked Potentials (MEP)
Description: This is a neurophysiological measure that determines the use of ipsilesional corticospinal tract. The paired-pulse TMS was applied at the respective hotspot for the elbow flexor muscle at the paretic arm over the ipsilesional primary motor cortex. The center of the coil was positioned tangentially to the skull. The patient was considered MEP+ if MEPs of any amplitude are observed at a consistent latency on at least 5 out 10 trials. After determining the status of MEP, at least eight more pulses were applied. We calculated average latency across all positive trials to determine the latency of MEP.
Time Frame: The latency of TMS-evoke MEP assessment is completed before and immediately after (within 30 min range) the intervention. The mean difference is then calculated (Post-Pre intevention) and recorded for each treatment group (anodal, cathodal, and sham).
Population: Eight subjects completed the study were analyzed.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Anodal Stimulation | Cathodal Stimulation | Sham
Number analyzed (Participants) | 8 | 8 | 8
ms | -24.21 (9.55) | -22.20 (10.10) | 1.16 (2.52)
Statistical Analysis 1: Comparison: Anodal Stimulation vs Cathodal Stimulation vs Sham; We compared anode to sham We compared cathode to sham We compared the change over time of anode to sham We compared the change over time of cathode to shal; Test type: Superiority; p = 0.0020, Regression, Cox — anode compared to sham p= 0.0020 cathode compared to sham p = 0.0088 anode over time anode compared to sham p <.0001 Cathode over time compared to sham p <.0001; Mean Difference (Final Values) = -24.2, 95% CI 2-sided [-32.2 to -16.2], Standard Deviation 9.5 — anode -24.2 (-32.2, -16.2) cathode -22.2 (-30.6, -13.8)

3. Other Pre Specified Outcome: Change in Brain Symmetry Index
Description: This is a neurophysiological measure used to quantify the symmetry or asymmetry between the left and right hemispheres of the brain. It was calculated using EEG data from a 3-minute resting state EEG recording. The scale of the index is from -1 to 1, where zero is considered perfect symmetry between hemispheres and values close to -1 and 1 indicate asymmetry.
Time Frame: The BSI assessment is completed before and immediately after (within 30 min range) the intervention. The mean difference is then calculated (Post-Pre intevention) and recorded for each treatment group (anodal, cathodal, and sham).
Population: 1 missing data for anodal and sham stimulation caused by a device failure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anodal Stimulation | Cathodal Stimulation | Sham
Number analyzed (Participants) | 7 | 8 | 7
score on a scale | 0.078 (0.077) | -0.068 (0.220) | -0.125 (0.213)
Statistical Analysis 1: Comparison: Anodal Stimulation vs Cathodal Stimulation vs Sham; e compare anode to sham We compare cathode to sham; Test type: Superiority; p = 0.0001, Regression, Linear — Compare anode to sham p= 0.0001 Compare cathode to sham p=0.1073 Compare anode change in time to sham p=0.0938 Compare cathode change in time to sham 0.0068; Using generalized estimating equations with group and time component; Mean Difference (Final Values) = 0.077, 95% CI 2-sided [0.00 to 0.10] — Anode = 0.077 (0.00, 0.10) Cathode = -.0.125 (-0.32 0.07 )

ADVERSE EVENTS:
Time Frame: 1 year, 3 months.
Arm/Group | Anodal Stimulation | Cathodal Stimulation | Sham
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT05174949/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT05174949/ICF_001.pdf